CLINICAL TRIAL: NCT02703532
Title: Evaluation of a CarePartner-Integrated Telehealth Rehabilitation Program for Persons With Stroke
Acronym: CARE-CITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); American Heart Association (Other)
Responsible Party: Principal Investigator, Sarah Blanton, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00070957; K23HD080837 (NIH)
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Stroke
Keywords: Therapy; Rehabilitation; Caregiver
MeSH Terms: conditions — Stroke | interventions — Constraint Induced Movement Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stroke Survivors with CARE-CITE Carepartners (Experimental): Stroke survivors with a carepartner randomized to the CARE-CITE intervention. Participants who have survived a stroke will receive constraint-induced movement therapy (CIMT) while their caregiver participates in an educational program.
  Interventions: Behavioral: Constraint-Induced Movement Therapy (CIMT)
- CARE-CITE Education Program Carepartners (Experimental): Caregivers (someone who assists in the care of stroke survivors) will participate in online CARE-CITE education while their partner (stroke survivor) receives therapy.
  Interventions: Behavioral: CARE-CITE Education Program
- Traditional Education Carepartners (Active Comparator): Caregivers (someone who assists in the care of stroke survivors) will participate in traditional education while their partner (stroke survivor) receives therapy.
  Interventions: Behavioral: Traditional Education
- Stroke Survivors with Traditional Education Carepartners (Active Comparator): Stroke survivors with a carepartner randomized to receive traditional education. Participants who have survived a stroke will receive constraint-induced movement therapy (CIMT) while their caregiver participates in an educational program.
  Interventions: Behavioral: Constraint-Induced Movement Therapy (CIMT)

INTERVENTIONS:
Behavioral: CARE-CITE Education Program — CARE-CITE is an online educational program developed to provide information that may help caregivers understand more about constraint-induced movement therapy (CIMT) and their potential roles in helping the stoke survivor gain as much benefit as possible from CIMT.
  If participants do not have access to a computer or tablet, they will be loaned an electronic tablet for the 2-3 week period of the study to access the information.
  Participants will be asked to review six educational modules over a period of 2-3 weeks while the stroke survivor receives CIMT.
  Participants will attend three in home evaluation visits; one at the beginning of the stroke survivors therapy sessions, one at the end of his/her therapy visit series, and a third evaluation one month later in which they will be asked to complete questionnaires. Evaluation visits will take approximately 1 ½ hours to complete.
  Arms: CARE-CITE Education Program Carepartners
Behavioral: Traditional Education — Investigators will explain constraint-induced movement therapy (CIMT) to caregivers and stroke survivors during the first home therapy session for the stroke survivor and provide traditional educational information about CIMT during therapy sessions as needed.
  Arms: Traditional Education Carepartners
Behavioral: Constraint-Induced Movement Therapy (CIMT) — Constraint-Induced Movement Therapy (CIMT) is one type of therapy that helps stroke survivors gain more use of their weaker arm.This therapy involves wearing a soft mitt (like a sock or oven mitt) on the stronger arm to remind the stroke survivor to use their weaker arm for daily activities and also intensive practice of tasks with the supervision of a therapist.
  Participants will attend three in home evaluation visits; one at the beginning of your therapy sessions, one at the end of your therapy visit series and a third evaluation one month later. These evaluation sessions will involve an evaluation of arm function and answering three questionnaires about how well the weaker arm works and how the stroke has affected daily activities. The interview questions and assessment will take approximately 1 ½ hours to complete.
  Arms: Stroke Survivors with CARE-CITE Carepartners; Stroke Survivors with Traditional Education Carepartners

SUMMARY:
The objective of this study is to identify the potential benefits of a home-based, intervention designed to facilitate carepartners' roles in stroke survivor rehabilitation. Stroke survivors and caregivers will participate in pairs. Stroke survivors will receive constraint induced movement therapy (CIMT). Caregivers of stroke survivors will be randomized to traditional caregiver education or a web based intervention for the duration of stroke survivor therapy. By learning the best way to involve family members in therapy, investigators hope to decrease the harmful effects of stroke.

DETAILED DESCRIPTION:
The objective of this study is to identify the potential benefits of a home-based, intervention designed to facilitate carepartners' roles in stroke survivor rehabilitation. Stroke survivors and caregivers will participate in pairs. Stroke survivors will receive constraint induced movement therapy (CIMT). Caregivers of stroke survivors will be randomized to traditional caregiver education or a web based intervention for the duration of stroke survivor therapy. A tablet will be provided to participants who do not have access to complete the web based intervention. All participants will be asked to complete questionnaires at the beginning of therapy, the end of therapy, and one month post therapy.

ELIGIBILITY:
Inclusion Criteria:

Stroke Survivors

* One month to five years post ischemic or hemorrhagic event
* Minimal to moderate upper extremity deficits (ability to initiate wrist and finger extension)
* Mini-mental screening test score of greater than 24
* Presence of a care partner

Caregivers

* At least 18 years old
* Ability to read and write English
* Mini-mental screening test score of greater than 24

Exclusion Criteria:

Stroke Survivors

* Severe cognitive deficits

Caregivers

* Significant cognitive deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-01; Primary Completion 2019-01-18 (Actual); Study Completion 2019-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Blanton, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Blanton S, Clark PC, Lyles RH, Cotsonis G, Jones BD, Reiss A, Wolf SL, Dunbar S. A web-based carepartner-integrated rehabilitation program for persons with stroke: study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2019 Apr 25;5:58. doi: 10.1186/s40814-019-0439-0. eCollection 2019. PMID 31057807

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant enrollment began in January 2016 and all study follow up was completed on January 8, 2019. Participants were enrolled at Emory University Hospital in Atlanta, Georgia.
Groups:
- CARE-CITE Education Program Carepartners: Carepartners (those assisting in the care of a stroke survivor) participated in online CARE-CITE education while their partner (the stroke survivor) received 10 sessions of constraint-induced movement therapy (CIMT).
- Traditional Education Carepartners: Carepartners (those assisting in the care of a stroke survivor) participated in traditional education while their partner (the stroke survivor) received 10 sessions of constraint-induced movement therapy (CIMT).
- Stroke Survivors With CARE-CITE Carepartners: Participants who have survived a stroke received 10 sessions of constraint-induced movement therapy (CIMT) while their carepartner participated in online CARE-CITE education.
- Stroke Survivors With Traditional Education Carepartners: Participants who have survived a stroke received 10 sessions of constraint-induced movement therapy (CIMT) while their carepartner participated in traditional education.
Period: Overall Study
Arm/Group | CARE-CITE Education Program Carepartners | Traditional Education Carepartners | Stroke Survivors With CARE-CITE Carepartners | Stroke Survivors With Traditional Education Carepartners
Started | 21 | 11 | 21 | 11
Completed | 19 | 10 | 19 | 10
Not Completed | 2 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Lost to Follow-up | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- CARE-CITE Education Program Carepartners: Carepartners (those assisting in the care of a stroke survivor) participated in online CARE-CITE education while their partner (the stroke survivor) received constraint-induced movement therapy (CIMT).
- Traditional Education Carepartners: Carepartners (those assisting in the care of a stroke survivor) participated in traditional education while their partner (the stroke survivor) received constraint-induced movement therapy (CIMT).
- Stroke Survivors With CARE-CITE Carepartners: Participants who have survived a stroke received constraint-induced movement therapy (CIMT) while their carepartner participated in online CARE-CITE education.
- Stroke Survivors With Traditional Education Carepartners: Participants who have survived a stroke received constraint-induced movement therapy (CIMT) while their carepartner participated in traditional education.
- Total: Total of all reporting groups
Arm/Group | CARE-CITE Education Program Carepartners | Traditional Education Carepartners | Stroke Survivors With CARE-CITE Carepartners | Stroke Survivors With Traditional Education Carepartners | Total
Number analyzed (Participants) | 21 | 11 | 21 | 11 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (12.6) | 60.1 (14.0) | 59.2 (15.3) | 63.3 (11.3) | 59.62 (13.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 6 | 9 | 5 | 34
  Male | 7 | 5 | 12 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 20 | 11 | 21 | 11 | 63
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 8 | 4 | 9 | 4 | 25
  White | 12 | 7 | 11 | 7 | 37
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 11 | 21 | 11 | 64

OUTCOME MEASURES:

1. Primary Outcome: Wolf Motor Function Test (WMFT)
Description: Motor ability and impairments will be assessed using the Wolf Motor Function Test (WMFT) an assessment tool used to evaluate upper extremity performance while providing insight into joint-specific and total limb movements. Values represent the amount of time, in seconds, to complete the assessment. Lower scores (faster speed) are indicative of higher functioning levels.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: This analysis includes stroke survivors completing the study visits; two carepartner and stroke survivor dyads in the CARE-CITE intervention were lost to follow-up between the end of treatment and the one month follow-up, and one dyad in the control group withdrew between the baseline visit and post-treatment visit.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Stroke Survivors With CARE-CITE Carepartners | Stroke Survivors With Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
seconds
  Baseline | 12.83 (2.27) | 9.38 (3.14)
  Post-treatment: number analyzed (Participants) | 21 | 10
  Post-treatment | 9.73 (2.27) | 4.70 (3.21)
  One Month Follow-up: number analyzed (Participants) | 19 | 10
  One Month Follow-up | 8.00 (2.32) | 5.18 (3.21)

2. Primary Outcome: Motor Activity Log (MAL) Score
Description: Upper extremity function and use will be assessed using the Motor Activity Log (MAL). The MAL is a semi-structured interview to assess arm function. Participants are asked to rate quality of movement (QOM) during 28 daily functional tasks. Items are scored on a 6-point ordinal scale, from 0 to 5, where 0 = the affected arm was of no use and 5 = affected arm is functioning normally. The total score is the average of all items and ranges from 0 to 5, where higher values indicate greater function of the arm that was impacted by the stroke.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stroke Survivors With CARE-CITE Carepartners | Stroke Survivors With Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 2.18 (0.18) | 2.34 (0.25)
  Post-treatment | 3.33 (0.18) | 3.59 (0.26)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 3.29 (0.19) | 3.39 (0.26)

3. Primary Outcome: Family Caregiver Conflict Scale (FCCS) Score
Description: Family conflict will be assessed using the Family Caregiver Conflict Scale (FCCS). The FCCS is 15-item scale that measures family conflict between caregivers and other family by assessing disagreements over caring for the care recipient with items such as: "We have disagreements when I ask family members to help me take care of our relative." Items are scored from 1 to 7 where 1 = not true at all and 7 = very true. total scores range from 15 to 105 and higher scores indicate greater family conflict.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: This analysis includes carepartners completing the study visits; two carepartner and stroke survivor dyads in the CARE-CITE intervention were lost to follow-up between the end of treatment and the one month follow-up, and one dyad in the control group withdrew between the baseline visit and post-treatment visit.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CARE-CITE Education Program Carepartners | Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 28.52 (2.24) | 20.00 (3.10)
  Post-treatment | 26.95 (2.24) | 21.87 (3.18)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 23.12 (2.30) | 18.57 (3.18)

4. Primary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D) Score
Description: Depressive symptoms among carepartners will be assessed by the Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D is a screening test for depression and depressive disorder. The CES-D measures the frequency and severity of 20 depressive symptoms experienced during the last week. Each item is scored from 0 to 3 where 0 = rarely and 3 = most days and certain items are reverse scored so that greater symptomatology is assigned a higher score. Total scores range from 0 to 60 and higher scores indicate greater symptoms of depression. Scores of 16 or greater are considered as an indicator of potential clinical depression.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CARE-CITE Education Program Carepartners | Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 8.33 (1.92) | 11.64 (2.65)
  Post-treatment | 8.14 (1.92) | 11.64 (2.72)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 7.84 (1.97) | 9.86 (2.72)

5. Secondary Outcome: Autonomy Support Family Care Climate Questionnaire for Stroke Survivor (FCCQ-SS) Score
Description: Autonomy support will be assessed using the Autonomy Support Family Care Climate Questionnaire for Stroke Survivor (FCCQ-SS). An autonomy supportive environment is characterized by empathy, communicating choice (avoiding controlling language), providing rationales and problem solving. Questions are asked about the stroke survivor's perspective on how much the carepartner provides an autonomy supportive environment for the stroke survivor. The FCCQ-SS includes 14 items scored from 1 to 7 where 1 = not true at all and 7 = very true. Item scores are averaged to provide an overall score between 1 and 7 where higher scores indicate the stroke survivor perceives receiving high autonomy support from the carepartner.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stroke Survivors With CARE-CITE Carepartners | Stroke Survivors With Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 6.36 (0.15) | 6.06 (0.20)
  Post-treatment | 6.39 (0.15) | 6.48 (0.20)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 6.54 (0.15) | 6.21 (0.20)

6. Secondary Outcome: Fugl-Meyer Assessment (FMA) Score
Description: Upper extremity impairment will be assessed by the Fugl-Meyer Assessment (FMA). The FMA includes 33 items that evaluate and measure recovery in post-stroke hemiplegic patients. Items are scored on a 3-point ordinal scale, from 0 to 2. Total scores range from 0 to 66 and higher scores indicates greater arm function.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stroke Survivors With CARE-CITE Carepartners | Stroke Survivors With Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 46.48 (1.80) | 49.91 (2.48)
  Post-treatment | 52.24 (1.80) | 53.36 (2.52)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 52.99 (1.81) | 55.46 (2.51)

7. Secondary Outcome: Confidence in Arm and Hand (CAHM) Scale Score
Description: Upper extremity self-efficacy will be assessed by the Confidence in Arm and Hand (CAHM) scale. The CAHM is a 20-item scale that examines self-efficacy for arm and hand function of the impaired upper extremity in individuals following stroke. Items are worded to assess task-specific self-confidence for unimanual and bilateral paretic arm and hand activities typically performed in home and community contexts. Items are scored on a scale of 0 (very uncertain) to 100 (very certain) and averaged to provide a total scale score ranging from 0 to 100. Higher scores indicate greater confidence with performing daily tasks with the impacted arm.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stroke Survivors With CARE-CITE Carepartners | Stroke Survivors With Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 58.45 (3.96) | 50.45 (5.47)
  Post-treatment | 74.12 (3.96) | 70.58 (5.64)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 76.76 (4.07) | 74.05 (5.64)

8. Secondary Outcome: Stroke Impact Scale (SIS) Score
Description: Quality of life will be assessed using the Stroke Impact Scale (SIS). The SIS is a stroke specific, self report questionnaire (59 items across 8 domains) that measures how a stroke has impacted a participant's health and life, including strength, memory and thinking, emotions and mood, communication, activities of daily living, mobility, function of affected upper extremity, and participation. Each item is rated in a 5-point Likert scale in terms of the difficulty the participant has experienced in completing each item. A score for each domain is obtained, ranging from 0 to 100 where higher scores indicate greater ability to perform tasks.
Time Frame: Baseline, 1 Month Post-treatment (up to Week 7)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Stroke Survivors With CARE-CITE Carepartners | Stroke Survivors With Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  SIS Strength - Baseline | 58.33 (3.26) | 51.14 (4.51)
  SIS Strength - 1 Month Post-treatment: number analyzed (Participants) | 19 | 10
  SIS Strength - 1 Month Post-treatment | 66.31 (3.37) | 70.17 (4.64)
  SIS Memory - Baseline | 84.01 (3.25) | 84.42 (4.49)
  SIS Memory - 1 Month Post-treatment: number analyzed (Participants) | 19 | 10
  SIS Memory - 1 Month Post-treatment | 88.09 (3.36) | 88.93 (4.64)
  SIS Mood - Baseline | 62.92 (2.72) | 62.63 (3.76)
  SIS Mood - 1 Month Post-treatment: number analyzed (Participants) | 19 | 10
  SIS Mood - 1 Month Post-treatment | 66.77 (2.81) | 69.04 (3.88)
  SIS Communication - Baseline | 92.52 (2.81) | 88.31 (3.88)
  SIS Communication - 1 Month Post-treatment: number analyzed (Participants) | 19 | 10
  SIS Communication - 1 Month Post-treatment | 92.61 (2.90) | 92.54 (4.01)
  SIS Activity - Baseline | 57.51 (2.40) | 54.73 (3.32)
  SIS Activity - 1 Month Post-treatment: number analyzed (Participants) | 19 | 10
  SIS Activity - 1 Month Post-treatment | 65.42 (2.46) | 61.71 (3.40)
  SIS Mobility - Baseline | 61.59 (2.97) | 52.93 (4.10)
  SIS Mobility - 1 Month Post-treatment: number analyzed (Participants) | 19 | 10
  SIS Mobility - 1 Month Post-treatment | 67.37 (3.04) | 58.65 (4.20)
  SIS Affected Arm - Baseline | 43.81 (3.75) | 34.55 (5.18)
  SIS Affected Arm - 1 Month Post-treatment: number analyzed (Participants) | 19 | 10
  SIS Affected Arm - 1 Month Post-treatment | 56.71 (3.86) | 53.43 (5.32)
  SIS Participation - Baseline | 43.45 (3.78) | 43.41 (5.23)
  SIS Participation - 1 Month Post-treatment: number analyzed (Participants) | 19 | 10
  SIS Participation - 1 Month Post-treatment | 53.50 (3.94) | 51.88 (5.43)

9. Secondary Outcome: Memory and Behavior Problems Checklist (MBPC) - Problem Frequency Score
Description: The MBPC is a 19-item caregiver-report instrument assessing observable behavioral problems in a loved one with dementia. Carepartners report how frequently problem behaviors occur on a scale from 0 to 4 where 0 = never occurs and 4 = occurs daily. Total scores range from 0 to 76, where higher scores indicate greater frequency of problematic behavior.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CARE-CITE Education Program Carepartners | Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 12.76 (2.39) | 21.91 (3.30)
  Post-treatment | 11.52 (2.39) | 16.63 (3.35)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 10.89 (2.42) | 14.03 (3.35)

10. Secondary Outcome: Autonomy Support Family Care Climate Questionnaire for Carepartner (FCCQ-CP) Scale Score
Description: Autonomy support for carepartners will be assessed by the Autonomy Support Family Care Climate Questionnaire for Carepartner (FCCQ-CP) Scale.An autonomy supportive environment is characterized by empathy, communicating choice (avoiding controlling language), providing rationales and problem solving. Questions are asked about the carepartner's perspective on how much they provide an autonomy supportive environment for the stroke survivor. The FCCQ-CP includes 14 items scored from 1 to 7 where 1 = not true at all and 7 = very true. Item scores are averaged to provide an overall score between 1 and 7 where higher scores indicate the carepartner thinks they are providing high autonomy support to the stroke survivor.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CARE-CITE Education Program Carepartners | Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 6.05 (1.97) | 6.21 (1.97)
  Post-treatment | 6.15 (1.97) | 6.27 (1.97)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 6.13 (1.97) | 6.15 (1.97)

11. Secondary Outcome: Piper Fatigue Scale (PFS) Score
Description: The Piper Fatigue Scale (PFS) is composed of 22 numerically scaled (0 to 10) items measuring four dimensions of subjective fatigue: behavioral/severity, affective meaning, sensory, and cognitive/mood. The total fatigue score is the average score for all questionnaire items and ranges from 0 to 10, where higher scores indicate greater fatigue.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CARE-CITE Education Program Carepartners | Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 3.82 (0.42) | 3.31 (0.58)
  Post-treatment | 2.69 (0.42) | 2.58 (0.60)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 2.97 (0.44) | 2.34 (0.60)

12. Secondary Outcome: Caregiver Strain Index (CSI) Score
Description: The CSI is a 12-question instrument measuring strain related to care provision. Carepartners respond to different statements with either "yes" or "no" where yes = 1 and no = 0. Total scores range from 0 to 12 with 0 indicating no caregiver strain and 12 indicating extreme strain. Positive responses to seven or more items on the index indicate a greater level of stress related to care giving.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CARE-CITE Education Program Carepartners | Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 5.52 (0.69) | 4.82 (0.96)
  Post-treatment | 5.00 (0.69) | 4.01 (0.98)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 3.78 (0.71) | 4.01 (0.98)

13. Secondary Outcome: Bakas Caregiving Outcomes Scale (BCOS) Score
Description: The BCOS is a 16-item scale asking about changes in the carepartner's social functioning, subjective well-being and physical health since they began caring for the stroke survivor. Participants responded to statements on a 7-point Likert scale (1=changed for the worst, 7=changed for the best). Total scores range from 16 to 112. Scores below 64 indicate that caring for the stroke survivor has resulted in negative changes, while scores above 64 indicate positive changes.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CARE-CITE Education Program Carepartners | Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 57.09 (2.63) | 55.91 (3.64)
  Post-treatment | 62.71 (2.63) | 59.56 (3.74)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 61.62 (2.70) | 60.62 (3.74)

14. Secondary Outcome: Caregiving Self Efficacy (Obtaining Respite Scale) Score
Description: The Caregiving Self Efficacy (Obtaining Respite Scale) measures the carepartner's self-efficacy for obtaining respite from caregiving. Five items are rated on a 0-100 scale where 0 = cannot do at all, 50 = moderately certain can do, and 100 = certain can do. A total score is obtained by averaging scores for the individual items. Total scores range from 0 to 100 with higher scores indicating that the carepartner has greater confidence in keeping up with their own activities while providing care to the stroke survivor.
Time Frame: Baseline, Post-treatment (up to Week 3), 1 Month Post-treatment (up to Week 7)
Population: as for outcome 3
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CARE-CITE Education Program Carepartners | Traditional Education Carepartners
Number analyzed (Participants) | 21 | 11
score on a scale
  Baseline | 66.44 (5.77) | 68.27 (7.97)
  Post-treatment | 69.52 (5.84) | 84.50 (8.20)
  1 Month Post-treatment Follow-up: number analyzed (Participants) | 19 | 10
  1 Month Post-treatment Follow-up | 71.80 (5.91) | 87.95 (8.20)

15. Secondary Outcome: Post Study System Usability Questionnaire (PSSUQ) Score
Description: The PSSUQ is a 19-item survey that measures users' perceived satisfaction with a product or system. Responses are given on a 7-point scale where 1 = strongly agree and 7 = strongly disagree. Responses are averaged to provide a total score between 1 and 7 where low answers indicate greater ease with using the CARE-CITE system.
Time Frame: Post-treatment (up to Week 3)
Population: This analysis includes carepartners who were in the CARE-CITE intervention study arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CARE-CITE Education Program Carepartners
Number analyzed (Participants) | 21
score on a scale | 1.48 (0.61)

ADVERSE EVENTS:
Time Frame: Adverse events related to the intervention were collected from the time of providing consent to participate in the study through the one month post-treatment study follow-up visit (approximately 7 weeks after the baseline assessment).
Arm/Group | CARE-CITE Education Program Carepartners | Traditional Education Carepartners | Stroke Survivors With CARE-CITE Carepartners | Stroke Survivors With Traditional Education Carepartners
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/11 | 0/21 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/11 | 0/21 | 1/11
Other Adverse Events (participants affected / at risk) | 0/21 | 0/11 | 9/21 | 3/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CARE-CITE Education Program Carepartners (N=21) | Traditional Education Carepartners (N=11) | Stroke Survivors With CARE-CITE Carepartners (N=21) | Stroke Survivors With Traditional Education Carepartners (N=11)
Lower extremity cellulitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — unrelated to the study intervention
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CARE-CITE Education Program Carepartners (N=21) | Traditional Education Carepartners (N=11) | Stroke Survivors With CARE-CITE Carepartners (N=21) | Stroke Survivors With Traditional Education Carepartners (N=11)
Fall (General disorders) | 0 | 0 | 7 | 2 — unrelated to study intervention
Heart rate increase (Vascular disorders) | 0 | 0 | 1 | 0 — unrelated to study intervention
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 — unrelated to study intervention
Muscle soreness or pain that limits participation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 — unrelated to study intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/32/NCT02703532/Prot_SAP_000.pdf